CLINICAL TRIAL: NCT06126822
Title: Safety and Immunogenicity of Ervebo® and Zabdeno® Booster Vaccines Against Ebola Virus Following Previous Vaccination with the Zabdeno/Mvabea® or Ervebo® Vaccine Schedules in DRC: a Mix-and-match Phase II RCT
Brief Title: Safety and Immunogenicity of Ervebo® and Zabdeno® Booster Vaccines Against Ebola Virus Following Previous Vaccination with the Zabdeno/Mvabea® or Ervebo® Vaccine Schedules in DRC
Acronym: EBO-BOOST
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Institute of Tropical Medicine, Belgium (Other)
Collaborators: Institut National pour la Recherche Biomedicale (INRB) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1706/23
Record Dates: First submitted 2023-10-05; First posted 2023-11-13 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Ebola Virus Disease
Keywords: Ebola vaccines
MeSH Terms: conditions — Hemorrhagic Fever, Ebola

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Zabdeno/Mvabea® vaccinated - Zabdeno® booster (Experimental): Participants previously vaccinated with the Zabdeno/Mvabea® vaccination schedule, will receive a single intramuscular Zabdeno® booster vaccine (0,5 ml) = homologous vaccination scheme.
  Interventions: Drug: Zabdeno® booster
- Zabdeno/Mvabea® vaccinated - Ervebo® booster (Experimental): Participants previously vaccinated with the Zabdeno/Mvabea® vaccination schedule, will receive a single intramuscular Ervebo® booster vaccine (1 ml) = heterologous vaccination scheme.
  Interventions: Drug: Ervebo® booster
- Ervebo® vaccinated - Ervebo® booster (Experimental): Participants previously vaccinated with Ervebo®, will receive a single intramuscular Ervebo® booster vaccine (1 ml) = homologous vaccination scheme.
  Interventions: Drug: Ervebo® booster
- Ervebo® vaccinated - Zabdeno® booster (Experimental): Participants previously vaccinated with Ervebo®, will receive a single intramuscular Zabdeno® booster vaccine (0,5 ml) = heterologous vaccination scheme.
  Interventions: Drug: Zabdeno® booster

INTERVENTIONS:
Drug: Zabdeno® booster — A single Zabdeno® booster vaccination
  Arms: Ervebo® vaccinated - Zabdeno® booster; Zabdeno/Mvabea® vaccinated - Zabdeno® booster
Drug: Ervebo® booster — A single Ervebo® booster vaccination
  Arms: Ervebo® vaccinated - Ervebo® booster; Zabdeno/Mvabea® vaccinated - Ervebo® booster

SUMMARY:
The goal of this randomized controlled trial is to investigate whether individuals in DRC previously vaccinated with Zabdeno/Mvabea® or Ervebo® vaccine schedules against Ebola virus can be safely and adequately boosted with homologous or heterologous vaccine schedules.

Participants will be randomized to receive either a homologous or heterologous vaccine schedule and will be asked to come to the clinic at prespecified timepoints over a period of 6 months to collect blood samples for comparison of immunological responses against Ebola virus between both schedules. Safety and tolerability of the vaccines will be evaluated by recording Adverse Events (AE's) and grading physical and vital signs evaluations.

DETAILED DESCRIPTION:
The aim of this randomized controlled with four arms is to investigate whether individuals previously vaccinated with Zabdeno/Mvabea® or Ervebo® vaccine schedules against Ebola virus can be safely and adequately boosted with homologous and heterologous vaccine schedules. We hypothesize that heterologous booster vaccine schedules generate a non-inferior boosting in antibodies and cellular responses against Ebola virus as compared to homologous schedules and incite a similar safety profile.

Based on the predefined variables (living place and time since vaccination), the research team will pre-select and re-contact individuals previously included in the Phase III EBOVAC vaccine database, EBOSURV participant database, and the Programme Élargi de Vaccination (PEV) database. Participants will be contacted by phone and, if they agree to participate, they are scheduled on predefined screening/recruitment days taken place at the 2 recruitment sites: INRB Goma and INRB Kinshasa.

A total of 624 participants will be included, 312 will be previously vaccinated with Zabdeno/Mvabea® and 312 participants with Ervebo®. Within those two groups, half of the participants (n=156) will be randomized to a single Ervebo® booster vaccine and the other half (n=156) to a single Zabdeno® booster vaccine. Participants will be asked to come to the clinic at prespecified timepoints over a period of 6 months to collect blood samples for comparison of antibody- and cellular response against EBOV between homologous and heterologous schedules. Safety and tolerability of the vaccines will be evaluated by recording Adverse Events (AE's) and grading physical and vital signs evaluations. An additional 50 non-vaccinated participants will be recruited in Kinshasa for assay optimization.

In case of insufficient participants living close to the recruitment centers, a community outreach will be undertaken with a lower amount of visits for logistical reasons.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who received either the Ervebo® vaccine (MSD), or the full Zabdeno, Mvabea® vaccine regimen (J&J) more than 4 months prior to recruitment
* Subjects between 18 and 50 years of age at time of randomization
* Subject must be willing and able to provide informed consent
* The subject must be in possession of an identification card (or other identification document)
* Agreement to refrain from blood donation and other vaccinations 30 days after booster vaccination
* Agreement to share and discuss participant's medical history, medical records and concomitant medications when relevant

Exclusion Criteria:

* Participants who previously experienced active Ebola Virus Disease (EVD)
* Receipt of any vaccine (licensed or experimental) within 30 days prior to recruitment
* Receipt of an additional booster dose of either Ervebo®, Zabdeno®, or any experimental Ebola vaccine
* Incorrect or incomplete primary vaccination scheme with the Zabdeno, Mvabea® (J&J) vaccine
* Administration of immunoglobulins and/or any blood products within three months prior to recruitment.
* Fever (>38°C) within last 24 hours prior to recruitment.
* Any confirmed or suspected immunosuppressive or immunodeficient state (incl. cancer and HIV); asplenia; recurrent severe infections and use of immunosuppressant medication within the last 6 months, except topical or short-term oral steroids.
* Severe and/or uncontrolled cardiovascular disease, respiratory disease, gastrointestinal disease, liver disease, renal disease, endocrine disorder and neurological illness (mild/moderate well controlled comorbidities are allowed)
* History of anaphylaxis, allergic disease or reactions to any component of the study vaccines
* History of bleeding disorder (e.g. factor deficiency, coagulopathy or platelet disorder), or prior history of significant bleeding or bruising following IM injections or venipuncture
* History of any thrombotic disorder, thrombocytopenia, thrombotic thrombocytopenia syndrome (TTP), or heparin-induced thrombocytopenia and thrombosis (HITT)
* Any other significant disease, disorder, planned surgery, or finding which may significantly affect the ability of the volunteer to participate in the study or impair interpretation of the study data
* Suspected or known alcohol or drug dependency
* Subject is not readily available by telephone, email or physical address

The non-vaccinated control group will also adhere to all the above in- and exclusion criteria, with exemption of:

* Agreement to refrain from blood donation and other vaccinations 30 days after study vaccination
* Subjects who received either the Ervebo® vaccine, or the full Zabdeno, Mvabea® vaccine regimen more than 4 months prior to recruitment

The latter is rather introduced as an additional exclusion criteria:

* Subjects who received either the Ervebo® vaccine or the full Zabdeno, Mvabea® vaccine regimen

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 624 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
To assess non-inferiority in EBOV-specific IgG levels elicited by a heterologous to a homologous booster vaccine schedule, by type of primary vaccination, 21 days after administration of the booster. | Day 21 after booster vaccination = Day 21
  FANG ELISA units/mL of anti-EBOV IgG

SECONDARY OUTCOMES:
To assess the safety of heterologous and homologous booster vaccine schedules, by type of primary vaccine schedule | Day 7, Day 21 and Month 6
  * The occurrence of solicited local Adverse Events (AEs) [Up to Day 7]
  * The occurrence of solicited systemic AEs [Up to Day 7]
  * The occurrence of unsolicited AEs [Up to Day 21]
  * The occurrence of Serious Adverse Events (SAE's) [Up to Month 6]
To compare the EBOV-specific IgG levels at D21 across all vaccine combinations | Day 21
  - FANG ELISA units/mL of anti-EBOV IgG at D21 after vaccination
To compare the fold change between D0 and D21 across all vaccine combinations | Day 0 and Day 21
  - Fold change in FANG ELISA units/mL of anti-EBOV IgG between D0 and D21
To compare the EBOV-specific binding and neutralizing antibodies to the glycoproteins of different EBOV variants across all vaccine combinations and timepoints | Day 0, Day 3, Day 7, Day 21, Month 6
  - The Mean Fluorescence Intensity (MFI) IgG levels against the GP variants [multiplexed Luminex assay - at D0, D3, D7, D21, M6]
To compare the EBOV-specific binding and neutralizing antibodies to the glycoproteins of different EBOV variants across all vaccine combinations and timepoints | Day 0, Day 21, Month 6
  - The 50% neutralizing titer (NT50) levels of the GP-specific antibodies [at D0, D21, M6]
To compare the EBOV-specific effector-memory T cell response across all vaccine combinations and timepoints | Day 0, Day 7, Day 21 and Month 6
  - The IFN-y, TNF-α and IL-2 Spot Forming Units (SFU) after T cell stimulation with GP peptide pools [at D0, D7, D21, M6]
To compare the EBOV-specific effector-memory B cell response across all vaccine combinations and timepoints | Day 0, Day 7, Day 21 and Month 6
  - The IgG1, IgG2, IgG3 Spot Forming Units (SFU) after B cell stimulation with recombinant GPs [at D0, D7, D21, M6]
To characterize the phenotype and polyfunctionality of the vaccine-induced T and B cell response by vaccine combination | at Day 0 and Day 21
  Proportions of EBOV GP-specific cell phenotypes and polyfunctional cells
To assess the impact of the participant age and sex on the vaccine-induced EBOV-specific bAbs | Day 21
  - FANG ELISA units/mL of anti-EBOV IgG at D21 after vaccination
To assess the impact of the participant age and sex on the vaccine-induced EBOV-specific bAbs | Day 0, Day 3, Day 7, Day 21 and Month 6
  - The Mean Fluorescence Intensity (MFI) IgG levels against the GP variants and VP40 [multiplexed Luminex assay - at D0, D3, D7, D21, M6]
To assess the impact of the participant age and sex on the vaccine-induced EBOV-specific nAbs | Day 0, Day 21 and Month 6
  - The 50% neutralizing titer (NT50) levels of the GP-specific antibodies [at D0, D21, M6]
To assess the impact of the participant age and sex on the vaccine-induced EBOV-specific T cells | Day 0, Day 7, Day 21 and Month 6
  - The IFN-y, TNF-α and IL-2 Spot Forming Units (SFU) after T cell stimulation with GP peptide pools [at D0, D7, D21, M6]
To assess the impact of the participant age and sex on the vaccine-induced EBOV-specific B cells | Day 0, Day 7, Day 21 and Month 6
  - The IgG1, IgG2, IgG3 Spot Forming Units (SFU) after B cell stimulation with recombinant GPs [at D0, D7, D21, M6]
To assess the impact of the participant age and sex on the vaccine-induced EBOV-specific T cells | Day 0, Day 21
  - Proportions of EBOV GP-specific cell phenotypes and polyfunctional cells [at D0, D21]

CONTACTS AND LOCATIONS:
Overall Officials: Wim Adriaensen, Prof., Principal Investigator — Institute of Tropical Medicine
Locations (2):
- Democratic Republic of the Congo (2):
  - Institut National de Recherche Biomédicale (INRB), Goma
  - Institut National de Recherche Biomédicale (INRB), Kinshasa

IPD SHARING:
Plan to Share IPD: No